CLINICAL TRIAL: NCT03352843
Title: Single Low-dose Primaquine Efficacy and Safety for Treatment of Uncomplicated Plasmodium Falciparum Malaria Based on Cytochrome P450 2D6 Activity in Bagamoyo District, Tanzania.
Brief Title: Single Low-dose Primaquine Efficacy and Safety.
Acronym: ESSLDPQP4502D6
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tropical Pesticides Research Institute, Tanzania (Other Government)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Principal Investigator, Richard Mwaiswelo, Research Scientist, Tropical Pesticides Research Institute, Tanzania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TMA2016CDF-1555
Record Dates: First submitted 2017-11-09; First posted 2017-11-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Primaquine — All patients will be administered with a single low-dose of primaquine in addition to standard artemether-lumefantrine regimen, and then followed-up for 28 days for clinical and laboratory assessment to assess safety and efficacy.

SUMMARY:
Background: The World Health Organization has recommended addition of a 0.25 mg/kg single-dose primaquine (PQ) to standard artemisinin-based combination therapy (ACT) for elimination of malaria in low transmission-settings and for containment in areas threatened by artemisinin resistance. However, PQ metabolism is dependent on a highly polymorphic cytochrome P450 (CYP) 2D6 isoenzyme which probably compromises the drugs' safety and efficacy, particularly in individuals with reduced isoenzyme activity. This trial therefore, aims to assess the safety and efficacy of 0.25 mg/kg single-dose PQ when added to standard artemether-lumefantrine regimen for clearance and sterilization of Plasmodium falciparum gametocytes in patients with CYP450 2D6 reduced/null activity as compared to those with normal/increased enzyme activity.

Methods: On hundred and fifty-five children aged between 1 and 10 years and with uncomplicated P. falciparum malaria will be enrolled, treated with standard artemether-lumefantrine regimen plus a 0.25 mg/kg single-dose of PQ and then followed up on days 0, 1, 2, 3, 7, 14, 21 and 28 for clinical and laboratory assessment. Primaquine will be administered together with the first dose of artemether-lumefantrine. Safety assessment will be performed using the Primaquine Roll Out Monitoring Pharmacovigilance Tool (PROMPT). Gametocytes will be detected and quantified by microscopy and Pfs25 mRNA quantitative nucleic acid sequence based amplification (QT-NASBA) on days 0 and 7. For a subset of 100 participants, post-treatment infectiousness will be assessed by mosquito feeding assays on day 7. The CYP2D6 status will be determined using a polymerase chain reaction (PCR) followed by a restriction fragment length polymorphism (RFLP). The primary outcome will be the safety of single low-dose primaquine in patients with CYP2D6 reduced/null compared to those with normal/increased activity.

Expected outcomes: The findings will provide the much-needed information on the safety and efficacy of single low-dose primaquine for clearance and sterilization of P. falciparum gametocytes in individuals with reduced/null compared to those with normal/increased CYP450 2D6 isoenzyme activity prior to the implementation of the treatment policy particularly in Africa.

ELIGIBILITY:
Inclusion Criteria:

* Age from 1 to 10 years
* Weight ≥ 10 kg
* Body temperature ≥ 37.5°C or history of fever in the last 24 hours
* Microscopy confirmed P. falciparum mono-infection
* Parasitemia level of 2000 - 200000/µL
* Ability to swallow oral medication
* Ability and willingness to abide by the study protocol and the stipulated follow up visits
* Written proxy informed consent from a parent/guardian.

Exclusion Criteria:

* Evidence of severe malaria or danger signs
* Known allergy to trial medicines
* Reported antimalarial intake ≤ 2 weeks
* Hemoglobin < 5 g/dL
* Blood transfusion within last 90 days
* Febrile condition other than malaria
* Known underlying chronic or severe disease

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Safety of single low-dose primaquine. | 6 months after the start of recruitment
  Proportion of participants with adverse and or serious adverse events between days 0 and 28 of follow up following treatment with a single low-dose primaquine in individuals with reduced/null compared to those with normal/increased CYP450 2D6 isoenzyme activity.

SECONDARY OUTCOMES:
Sterilization of gametocytes | 6 months after the start of recruitment
  Proportion of participants with infected mosquitoes following membrane feeding experiment on day 7.
Gametocytes carriage on day 7 | 12 months after the start of recruitment
  Proportion of participants with gametocytes carriage measured by QT-NASBA on day 7

CONTACTS AND LOCATIONS:
Overall Officials: Richard O Mwaiswelo, PhD, Principal Investigator — Tropical Pesticides Research Institute
Locations (1):
- Tropical Pesticides Research Institute (TPRI), Arusha, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Shared after the primary findings have been published
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Mwaiswelo RO, Ngasala B, Msolo D, Kweka E, Mmbando BP, Martensson A. A single low dose of primaquine is safe and sufficient to reduce transmission of Plasmodium falciparum gametocytes regardless of cytochrome P450 2D6 enzyme activity in Bagamoyo district, Tanzania. Malar J. 2022 Mar 12;21(1):84. doi: 10.1186/s12936-022-04100-1. PMID 35279143